CLINICAL TRIAL: NCT07352904
Title: Exploration Strategies in Night Vision Sensors
Acronym: STRAT-JVN
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00047-42
Record Dates: First submitted 2025-09-18; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity
Keywords: visual strategy; Night Vision Goggles; eyetracking; visual fatigue
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this clinical trial is to identify a variation in visual strategy characterized by both head movements and eye movements of healthy volunteers during a target detection task when images simulating night vision goggles (NVG) are presented, compared to a situation in which the images simulate a natural environment.

To highlight changes in environmental scanning with simulated images from NVG, objective measurements will be collected:

* eye movements characterized by saccades (speed, latency, and number) for each stimulus
* head movements (horizontal angle of the participant's head) for each stimulus and throughout the exposure

Participants sit facing a screen (9.90 m x 2.10 m) onto which a virtual scene is projected. The objective is to correctly identify, as quickly as possible, a target stimulus (represented by a tank) that may appear in the scene. They must use the directional arrows on a game controller to indicate whether the tank is moving to the left or to the right.

There are four visits involving four viewing conditions in which the task remains the same:

* With restricted field of view and a normal scene.
* Without restricted field of view and a scene simulating the vision obtained by NVGs.
* With restricted field of view and a scene simulating the vision obtained by NVGs.
* Without restricted field of view and a normal scene. Regarding the content of the scene, half of the tests in each visit involve a so-called poor scene when fog is simulated, or an enriched scene when there is no fog. Each visit lasts approximately one hour and thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with social security;
* Normal vision or vision corrected with lenses (far vision ≤ 0.03 log unit (≥ 9/10) OD/OG/binocular);
* No current or past ocular or binocular pathology: strabismus or amblyopia;
* Signed non-objection form.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Incapacitated adults;
* Individuals who do not understand French (written or spoken).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French volunteers
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Eye movements characterized by saccades (speed, latency, and number) for each stimulus | Day 1 (Visit 1) and during follow-up visits at Day 2 (Visit 2), Day 3 (Visit 3), and Day 4 (Visit 4)
  Measurements from eyetracker
Head movements (horizontal angle of the participant's head) for each stimulus and throughout the exposure | Day 1 (Visit 1) and during follow-up visits at Day 2 (Visit 2), Day 3 (Visit 3), and Day 4 (Visit 4)
  Measurements extract from motion capture

SECONDARY OUTCOMES:
The average stimulus detection times. | Day 1 (Visit 1) and during follow-up visits at Day 2 (Visit 2), Day 3 (Visit 3), and Day 4 (Visit 4)
  Measurements from an eyetracker
Number of correct responses to the perceptual task | Day 1 (Visit 1) and during follow-up visits at Day 2 (Visit 2), Day 3 (Visit 3), and Day 4 (Visit 4)
  Extract with software
Visual fatigue will be measured using a questionnaire | Day 1 (Visit 1) and during follow-up visits at Day 2 (Visit 2), Day 3 (Visit 3), and Day 4 (Visit 4)
  To highlight subjective visual fatigue generated by changes in visual search strategies using simulated images from night vision sensors.